CLINICAL TRIAL: NCT02353533
Title: Endoscopic Full-thickness REsection of Residual Colorectal Lesions - The FiRE Study
Acronym: FiRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Peter Klare, Dr. med. Peter Klare, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FiRE
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Adenoma
Keywords: adenoma; EMR; FTRD; non- lifting; colon
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMR (Other): Standard EMR technique
  Interventions: Device: EMR
- FTRD (Experimental)
  Interventions: Device: over- the- scope full- thickness resection device (FTRD)

INTERVENTIONS:
Device: over- the- scope full- thickness resection device (FTRD) — Endoscopic resection of adenomatous lesions of the colon using the over- the- scope full- thickness resection device
  Arms: FTRD
Device: EMR — Standard endoscopic mucosal resection using a resection snare
  Arms: EMR

SUMMARY:
Adenomatous lesions of the colon are premalignant lesions which have the potential to develop cancer. Therefore adenomas should be resected endoscopically (endo- mucosa resection, EMR). EMR is conducted after submucosal injection of saline which allows to lift the desired lesion prior to resection. In some cases EMR is complicated due to incomplete or failed lifting after the injection of saline. This so- called "non- lifting" sign is a predictor for malignancy of the lesion. Difficult- to- lift polyps are also difficult- to- resect. A higher proportion of these lesions fail to be resected completely using the EMR technique.

Alternatively, an over- the- scope full- thickness resection device (FTRD) can be used in order to resect colonic lesions. The FTRD technique has been described elsewhere (Schmidt et al. Gastroenterology 2014; 147: 740-742.e2). No comparative data exists until now on the performance of FTRD resection compared to standard EMR resection of difficult- to- resect colon adenomas.

In this study the investigators aim to compare the success of FTRD versus EMR of difficult- to- resect adenomatous lesions (≤ 20 mm).

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years
* adenomatous lesion 10-20 mm in size with expected difficulties regarding EMR (e.g. "non- lifting sign")

Exclusion Criteria:

* patients < 18 years
* lesions > 20 mm in size
* high risk carcinomas ("deep submucosal carcinoma")
* American Society of Anesthesiologists (ASA) class IV and higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Success of resection | 3 month
  Success of resection: Complete resection (R0) according to clinical and/or histopathological assessment

SECONDARY OUTCOMES:
Duration of procedure | up to 1 day (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan von Delius, MD, Study Director — II. Medizinische Klinik, Klinikum rechts der Isar der Technischen Universität München, Germany
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Germany